CLINICAL TRIAL: NCT03602872
Title: Phase I, Open Label Study to Assess the Safety and Tolerance of a Single Intraarticular Dose of STEMEDICA's Human Allogeneic Bone Marrow Derived Mesenchymal Stem Cells, in Subjects With Knee Osteoarthritis.
Brief Title: Safety of Allogeneic Bone Marrow Derived Mesenchymal Stem Cells in Subjects With Osteoarthritis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor to start with different protocol, postponed due to COVID
Sponsor: Clinica Santa Clarita, Mexico (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO-OAR-BW-001
Record Dates: First submitted 2018-07-17; First posted 2018-07-27 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis, safety, MSCs
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1 (Experimental): Subjects will receive a single intraarticular 20x10^6 dose of Human allogeneic mesenchymal bone marrow derived stem cells, in the most symptomatic target (knee) joint.
  Interventions: Biological: Human allogeneic mesenchymal bone marrow derived stem cells
- Group 2 (Experimental): Subjects will receive a single intraarticular 20x10^6 dose of Human allogeneic mesenchymal bone marrow derived stem cells, in the most symptomatic target (knee) joint.
  Interventions: Biological: Human allogeneic mesenchymal bone marrow derived stem cells
- Group 3 (Experimental): Subjects will receive a single intraarticular 20x10^6 dose of Human allogeneic mesenchymal bone marrow derived stem cells, in the most symptomatic target (knee) joint.
  Interventions: Biological: Human allogeneic mesenchymal bone marrow derived stem cells

INTERVENTIONS:
Biological: Human allogeneic mesenchymal bone marrow derived stem cells — Intraarticular administration of 20x10^6 MSCs

SUMMARY:
The aim of this study is to assess the safety of Stemedica's mesenchymal stem cells in patients with knee osteoarthritis. The route of administration is intraarticular. Safety will be evaluated by AE/SAE incidence and administration tolerance. The subjects will undergo follow-up for 52 weeks. The target population is subjects with knee osteoarthritis (grade II-III in Kellgren-Lawrence scale).

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers between 35-65 years.
* X-ray evidence of osteoarthritis (grade II-III in Kellgren-Lawrence).
* Chronic joint pain (>5 visual analogue scale) in knee.
* BMI ≤ 29.
* Voluntary acceptance and signature of informed consent.
* Willing to attend study visits and lab sample recollection.
* Lab values within normal reference values.
* Willing to use effective birth control methods.

Exclusion Criteria:

* Inflammatory arthritis.
* Generalized infection.
* Active cancer or history of cancer in the past 5 years.
* Receiving oral or intraarticular steroids.
* Positive labs for HIV, Hepatitis B or C.
* Recent trauma in the target joint.
* Debris in joint.
* Subjects that have undergone or need to undergo arthroscopic knee surgery in the target joint.
* History of joint substitution, intraarticular fractures, osteotomy, arthroplasty or menisectomy.
* Clinically significant knee misalignment.
* Other illnesses that the investigator considers clinically significant.
* Participating in another clinical trial three months before enrolling.
* Women that are pregnant, lactating or result positive in the pregnancy test during screening.
* Known allergies to bovine products.
* Subjects taking anticoagulants.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation of all AE/SAEs | From the first dosing of the first subject up to 30 days after the last follow up of the last dosed subject
  All AE/SAE will be assessed for causality and reported utilizing MedDRA terminology.

SECONDARY OUTCOMES:
Procedure tolerance (procedure pain/discomfort incidence) | 7 days after subject receives dosing
  The procedure tolerance will be evaluated through a questionnaire for procedure pain/discomfort incidence.
WOMAC questionnaire | From the first dosing of the first subject up to 30 days after the last follow up of the last dosed subject
  The WOMAC questionnaire will be used to evaluate any preliminary efficacy findings throughout the study completion.
OAKHQOL questionnaire | From the first dosing of the first subject up to 30 days after the last follow up of the last dosed subject
  The OAKHQOL questionnaire will be used to evaluate any preliminary efficacy findings throughout the study completion.

CONTACTS AND LOCATIONS:
Overall Officials: José F Izquierdo, M.D., Principal Investigator — External
Locations (1):
- Clinica Santa Clarita, Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: No